CLINICAL TRIAL: NCT03445858
Title: A Pilot Study of Pembrolizumab in Combination With Decitabine and Hypofractionated Index Lesion Radiation in Pediatric and Young Adult Patients With Relapsed and Refractory Solid Tumors or Lymphoma
Brief Title: Pembrolizumab in Combination With Decitabine and Hypofractionated Index Lesion Radiation in Pediatrics and Young Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pembro_BT_1603
Record Dates: First submitted 2018-02-14; First posted 2018-02-26 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Childhood Solid Tumor; Childhood Lymphoma; Relapsed Cancer; Refractory Cancer; Adult Solid Tumor; Adult Lymphoma
Keywords: Pediatric; Immunotherapy; Radiation; Radiotherapy; PD-1; Decitabine; DNMT; Epigenetic; Solid Tumor; Saroma; Lymphoma; Checkpoint; Abscopal; Cancer; Immune; SBRT
MeSH Terms: conditions — Recurrence; Neoplasms; Lymphoma | interventions — pembrolizumab; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab, Decitabine, Radiation (Experimental): Patients will receive pembrolizumab and decitabine every 28 days, and a single 3 day course of fixed-dose hypofractionated radiotherapy to one or more index lesions.
  Interventions: Drug: Pembrolizumab; Drug: Decitabine; Radiation: Hypofractionated Index Site Radiation

INTERVENTIONS:
Drug: Pembrolizumab — Patients will receive pembrolizumab every 28 days.One cycle lasts 28 days. Cycles may repeat for a total of 26 cycles if patient meets criteria to continue protocol therapy.
  Other Names: Keytruda
Drug: Decitabine — Patients will receive decitabine every 28 days.One cycle lasts 28 days. Cycles may repeat for a total of 26 cycles if patient meets criteria to continue protocol therapy.
  Other Names: Dacogen
Radiation: Hypofractionated Index Site Radiation — Patients will receive a single 3 day course of fixed-dose hypofractionated radiotherapy to one or more index lesions during the first cycle only.

SUMMARY:
This pilot study is designed to assess the safety, tolerability, and preliminary anti-tumor activity of the combination of pembrolizumab, decitabine and fixed-dose hypofractionated index site radiotherapy in pediatric and young adult patients with relapsed, refractory or progressive non-primary CNS solid tumors and lymphomas.

Primary Objectives

* To determine the feasibility of administering pembrolizumab in combination with decitabine and hypofractionated index lesion radiation
* To identify the treatment related toxicity and tolerability of the combination of decitabine and pembrolizumab with hypofractionated index lesion radiation

Secondary Objective

To preliminarily define the anti-tumor efficacy of the combination of pembrolizumab, decitabine and hypofractionated index lesion radiation in patients with relapsed, refractory, or progressive non-CNS solid tumors and lymphomas using overall response rate (CR + PR) by irRECIST after 2 cycles of therapy.

Exploratory Objectives

To profile the kinetics of the immune response and to correlate with promotor methylation changes, nuclear imaging, stool microbiota diversity, and tumor associated antigen immune responses.

DETAILED DESCRIPTION:
Patients will receive pembrolizumab and decitabine every 28 days, and a single 3 day course of fixed-dose hypofractionated index site radiotherapy to one or more index lesions.

One cycle lasts 28 days. Radiation is given in Cycle 1 only. Cycles may repeat for a total of 26 cycles if patient meets criteria to continue protocol therapy.

ELIGIBILITY:
Criteria: Inclusion Criteria:

* Age: greater than or equal to 12 months and less than or equal to 40 years.
* Diagnosis: Patients must have had histologic verification of malignancy at original diagnosis or relapse. Eligible diagnoses include:

  * Relapsed or refractory solid tumors (excluding primary CNS tumors)
  * Lymphoma in second or greater relapse or with refractory disease
* Disease Evaluation: Patients must have evaluable or measurable disease (patients with evaluable disease must have at least one lesion that is amenable to radiation as below).
* Patients with stable non-brainstem CNS metastases may be eligible.
* Therapeutic Options: Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life.
* Performance Level: Lansky/Karnofsky greater than or equal to 50.
* Prior Therapy: Patients who have previously received inhibitors of PD-1, PD-L1, CTLA4 or other immune checkpoint inhibitors, regardless of response, are eligible as long as they had not experienced a medically significant immune related adverse event that required treatment with supraphysiologic steroids or other immunomodulatory drug.
* Patients must have recovered from the acute toxic effects of all prior anti-cancer chemotherapy and meet the following:

  * Myelosuppressive chemotherapy: At least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea).
  * Hematopoietic growth factors: At least 21 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor.
  * Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent.
  * Immunotherapy: At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines.
  * Monoclonal antibodies: At least 4 weeks after the last dose of a monoclonal antibody.
  * XRT: At least 14 days after local palliative XRT (limited field); At least 150 days must have elapsed if prior TBI, craniospinal XRT or radiation treatment resulting in greater than or equal to 50% of the pelvis receiving greater than or equal to 10 Gy.
  * Stem Cell Infusion without TBI: At least 84 days must have elapsed after autologous stem cell transplant or stem cell infusion. Patients having received allogeneic stem cells within the past 5 years are not eligible.
* Adequate Bone Marrow Function Defined as:

  * Peripheral absolute neutrophil count (ANC) greater than or equal to 750/mm3
  * Platelet count greater than or equal to 75,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
  * Hemoglobin greater than or equal to 8 (transfusions allowed)
  * Patients with known bone marrow involvement will no longer be eligible for this study.
* Adequate Renal Function Defined as:

  o Creatinine clearance, cystatin C based GFR, or radioisotope GFR greater than or equal to 70ml/min/1.73 m2 or a serum creatinine based on protocol requirements.
* Adequate Liver Function Defined as:

  * Direct bilirubin less than or equal to 1.5 x upper limit of normal (ULN) for age
  * SGPT (ALT) less than or equal to 3.0 x upper limit of normal (ULN). For patients with known liver metastases or primary tumor, SGPT (ALT) less than or equal to 5 x upper limit of normal (ULN) may be accepted. For the purposes of this study, the ULN of SGPT is 45 U/L.
* Adequate Cardiac Function Defined as:

  * Ejection fraction of greater than or equal to 50% by echocardiogram (3D if available) or cardiac MRI.
  * QTC less than or equal to 480 msec.
* Adequate Pulmonary Function Defined as:

  o Pulse oximetry greater than 94% on room air and no dyspnea at rest.
* Radiation Considerations:

  * Patients must have at least one non-CNS lesion amenable to radiation as defined in the protocol and at the discretion of the Study Chair.
  * Patients with previously irradiated sites of disease may be considered eligible if potential index lesions meet the following: There has been documented progression at that site (by RECIST or for neuroblastoma patients enrolled with evaluable disease, persistent MIBG avidity), and Re-irradiation would not expose the patient to a substantial increase in toxicity (as determined by consultation with co-principal investigator or designee and treating oncologist).

Exclusion Criteria:

* Patients with primary CNS tumors, brainstem metastases, and/or carcinomatous meningitis are not eligible.
* Pregnant or breast-feeding women will not be entered on this study.
* Corticosteroids and other immunosuppressive therapy: Patients requiring systemic corticosteroids or other immunosuppressive medication within 7 days prior to enrollment are not eligible with the exception of physiologic replacement doses of corticosteroids.
* Patients who are currently receiving another investigational drug are not eligible.
* Patients who are currently receiving other anti-cancer agents are not eligible.
* Patients with a history of a non-thyroiditis autoimmune disorder are not eligible. Asymptomatic laboratory abnormalities (e.g. ANA, rheumatoid factor) will not render a patient ineligible in the absence of a diagnosis of an autoimmune disorder. Autoimmune thyroiditis will not render a patient ineligible.
* Patients with known hepatitis B (HBsAg reactive) or C (HCV RNA -qualitative is detected) are excluded.
* Patients with HIV are excluded if they have detectable viral loads or CD4 count is below 400 or they are not compliant with antiretroviral agents.
* Patients who have an uncontrolled infection are not eligible.
* Patients with immunodeficiency syndromes are not eligible.
* Patients with a history of clinically significant cardiac disease are not eligible.
* Patients with ongoing interstitial lung disease or pneumonitis are not eligible.
* Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction).
* Patients who have received a live vaccine less than or equal to 30 days prior to enrollment are ineligible.
* Patients who have received a prior solid organ transplant at any time, or allogeneic bone marrow transplantation within the past 5 years (or have signs or symptoms of GVHD) are not eligible.

Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

Ages: 12 Months to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of administering Pembrolizumab in combination with Decitabine and hypofractionated index radiation | Days 1 thru 57
  Incidence of number of patients who experience a DLT

SECONDARY OUTCOMES:
Identification of treatment related toxicities and tolerability | Days 1 thru 57
  Incidence of adverse events (toxicities) according to NCI CTCAE version 5.0
Define anti-tumor efficacy of treatment combination of pembrolizumab, decitabine, and hypofractionated index radiation (per irRECIST criteria) | 2 cycles (56 days)
  Incidence of patients who experience an overall complete response or partial response to study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Brian Turpin, DO, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States